CLINICAL TRIAL: NCT06487312
Title: Clinical Application of Multi-organ Multi-task Autonomous Ultrasound Embodied Intelligent Robot
Brief Title: Clinical Trial to Evaluate the Effectiveness and Safety of a Remote Automated Ultrasound Diagnostic System for Automated Ultrasound Examinations: a Prospective, Multicenter Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Xin-Wu Cui, Professor, Tongji Hospital
Other Study IDs: 2024S730
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Ultrasound; Thyroid; Carotid Artery; Liver; Gallbladder; Spleen; Pancreas; Kidney
Keywords: Ultrasound Intelligent Robot; Multitasking; Automated Ultrasound; Clinical application
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Age ≥ 18 years old, regardless of gender, who need ultrasound examination; 3) Voluntarily participat
  Interventions: Device: Test equipment: Name: Remote automatic ultrasound diagnostic system (Wuhan Cooper Technology Co., Ltd.) Model: CORUS-A30

INTERVENTIONS:
Device: Test equipment: Name: Remote automatic ultrasound diagnostic system (Wuhan Cooper Technology Co., Ltd.) Model: CORUS-A30 — A clinical trial to evaluate the effectiveness and safety of a remote automated ultrasound diagnostic system for automated ultrasound examination using a remote automated ultrasound diagnostic system (model: CORUS-A30, Wuhan Cooper Technology Co., Ltd., China).

SUMMARY:
The purpose of this clinical trial is to verify the safety and effectiveness of the remote automatic ultrasound diagnosis system produced by Wuhan Cooper Technology Co., Ltd. for automatic ultrasound examination. It aims to answer the main questions:

Can the robot complete automatic ultrasound scanning of multiple systems and organs such as liver, gallbladder, spleen, pancreas, kidney, thyroid, carotid artery, etc.? Will there be medical safety issues during the robot's scanning process?

ELIGIBILITY:
Inclusion Criteria:

* 1) Aged ≥ 18 years old, regardless of gender; 2) Those who need to undergo ultrasound examination; 3) Those who voluntarily participate in this trial and sign the informed consent form.

Exclusion Criteria:

* 1) Those who are allergic to ultrasound coupling agents; 2) Those who are unable to undergo long-term ultrasound examinations due to physical or mental reasons (such as intellectual disability, mental illness, etc.); 3) Those who have suffered severe trauma or burns within the past month; 4) Pregnant or breastfeeding women; 5) Those who have participated in other clinical trials within the past month; 6) Other subjects deemed by the researchers to be unsuitable for participating in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will recruit adults over 18 years old, especially those who need multi-organ ultrasound examinations. Participants need to be able to understand and sign the informed consent. We hope to include patients of different ages, genders, and health conditions to ensure the wide applicability of the study results. Your participation will help us test and improve the autonomous ultrasound robot so that it can work effectively in a variety of populations.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Image scanning pass rate | 12 months
  Each subject is subjected to ultrasound examination using the corresponding probe using the test device. The image quality of each part is evaluated according to the examination site and the image evaluation standards of each part (see Appendix 1); whether it meets the doctor's diagnostic needs is determined according to the scan completeness evaluation standards (see Appendix 2). The examination sites include: abdomen (liver, gallbladder, pancreas, spleen and kidney), superficial small organs (thyroid) and peripheral blood vessels (carotid artery). Each subject can undergo examination of all parts or some parts on the same day. If the subject has a history of organ resection surgery, ultrasound examination of the corresponding part will not be performed. The expert group consists of three researchers. The three expert group researchers evaluate the ultrasound image video and standard cross-section diagram collected by the test device back to back. When the results are inconsistent, t

CONTACTS AND LOCATIONS:
Locations (1):
- Xin-Wu Cui, Wuhan, Hubei, China